CLINICAL TRIAL: NCT04293822
Title: Topical Cetirizine Gel Versus Minoxidil 5% Gel in Treatment of Androgenetic Alopecia
Brief Title: Topical Cetirizine 1% vs Minoxidil 5% Gel in Treatment of Androgenetic Alopecia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Abdalla Ibrahim, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AssiutU Dermatology
Record Dates: First submitted 2020-02-21; First posted 2020-03-03 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Cetirizine; Gels; Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patients will be randomly divided into 2 groups; each group contains 30 patients. Patients in both groups will be given the treatment in identical non-labeled bottles with a code and neither the patient nor the doctor will know which treatment is given and what the code referred to. The patients will be instructed to use the treatment twice daily for 6 month duration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study group (Experimental): Group of 30 patients randomly selected will use topical Cetirizine 1% gel twice daily over a period of 6 months, where the treatment will be given in identical non-labeled bottles with a code and neither the patients, healthcare provider nor the investigator will know which treatment is given and what the code referred to.
  Interventions: Drug: Cetirizine
- Control group (Active Comparator): Group of 30 patients randomly selected will use topical Minoxil 5% gel twice daily over a period of 6 months, where the treatment will be given in identical non-labeled bottles with a code and neither the patients, healthcare provider nor the investigator will know which treatment is given and what the code referred to.
  Interventions: Drug: Minoxidil

INTERVENTIONS:
Drug: Cetirizine — The patients will be randomly divided into 2 groups; each group contains 30 patients. Patients in both groups will be given the treatment in identical non-labeled bottles with a code and neither the patient nor the doctor will know which treatment is given and what the code referred to. The patients will be instructed to use the treatment twice daily for 6 month duration.
  This group will use Cetrizine 1% gel, which will be prepared at the department of Pharmaceutics, Faculty of Pharmacy, Assiut University in the form of Nano-transferosomes (NTF).
  Other Names: Cetirizine 1% Gel
  Arms: Study group
Drug: Minoxidil — The patients will be randomly divided into 2 groups; each group contains 30 patients. Patients in both groups will be given the treatment in identical non-labeled bottles with a code and neither the patient nor the doctor will know which treatment is given and what the code referred to. The patients will be instructed to use the treatment twice daily for 6 month duration.
  This group will use Minoxidil 5% gel
  Other Names: Minoxidil 5% Placebo
  Arms: Control group

SUMMARY:
Androgenetic alopecia (AGA), also known as androgenic alopecia or male pattern baldness, is the most common type of progressive hair loss. It is a polygenetic condition with variable degree of severity, age of onset, and location of hair loss.

Male AGA (MAGA) is clearly an androgen-dependent condition and, although the mode of inheritance is uncertain, a genetic predisposition is observed.

Regarding treatment of AGA; in most cases it's challenging and unsatisfactory. Finasteride and Minoxidil 2-5 % solution are the only US Food and Drug Administration (FDA) approved treatment options for MAGA.

On the basis of hypertrichosis observed in patients treated with analogues of prostaglandin PGF2a (i.e. latanoprost used for glaucoma), it was supposed that prostaglandins would have an important role in the hair growth (Nieves et al., 2014).

Multiple studies had claimed that prostaglandins are deregulated in both alopecia areata (AA) and AGA.

Cetirizine, is a safe and selective second-generation histamine H1 receptor antagonist widely used. It has anti-inflammatory properties. Studies have shown cetirizine causes a significant reduction in both the inflammatory cell infiltrate and PGD2 production.

The oral administration of cetirizine is commonly leads to different systemic side effects. Thus the topical formulation is expected to be an effective tool for avoiding the oral side effects as well as better targeting, but unfortunately, no topical formulation of cetirizine is available in the market till date.

DETAILED DESCRIPTION:
Androgenetic alopecia (AGA), also known as androgenic alopecia or male pattern baldness, is the most common type of progressive hair loss. It is a polygenetic condition with variable degree of severity, age of onset, and location of hair loss.

Hair loss typically begins with bi-temporal recession of the frontal hairline, followed by diffuse hair thinning at the vertex, and eventual complete loss of hair at the center of the vertex. The bald patch at the vertex subsequently joins the frontal receding hairline, leaving an island of hair on the frontal scalp, which finally disappears leaving hair only in the parietal and occipital zones producing the characteristic "horseshoe" pattern.

Androgenetic alopecia is classified according to the Hamilton-Norwood scale into grades (from I to VII).

AGA features a progressive miniaturization of the hair follicle leading to vellus transformation of terminal hair which results from an alteration in hair cycle dynamics: anagen phase duration gradually decreases and that of the telogen phase increases. As the anagen phase duration determines hair length, the new anagen hair becomes shorter, eventually leading to bald appearance.

The etiology of AGA is multifactorial and polygenetic. Male AGA (MAGA) is clearly an androgen-dependent condition and, although the mode of inheritance is uncertain, a genetic predisposition is observed, while in female AGA (FAGA) the role of androgens is still uncertain.

Regarding treatment of AGA; in most cases it's challenging and unsatisfactory. Finasteride and Minoxidil 2-5 % solution are the only US Food and Drug Administration (FDA) approved treatment options for MAGA.

Finasteride is a type 2 5α-reductase inhibitor that decreases the conversion of testosterone to dihydrotestosterone (DHT), which is responsible for the miniaturization of the hair follicle seen in MAGA.

Minoxidil is a direct arteriolar vasodilator acts by opening potassium channels. Unwanted hair growth was observed as an adverse effect in 24-100 % of patients treated by Minoxidil for hypertension. Minoxidil 2 % solution was approved in 1988, while the 5 % solution was approved in 1991, and the 5 % foam in 2016 for MAGA.

On the basis of hypertrichosis observed in patients treated with analogues of prostaglandin PGF2a (i.e. latanoprost used for glaucoma), it was supposed that prostaglandins would have an important role in the hair growth.

Their action is variable depending on the class they belong to: PGE and PGF2a play a generally positive role on the hair growth, while PGD2 an inhibitory role on the hair growth.

Multiple studies had claimed that prostaglandins are deregulated in both alopecia areata (AA) and AGA.

Garza in 2012 found elevated levels of prostaglandin D2 synthase (PTGDS) at the mRNA and protein levels in bald scalp versus haired scalp of men with AGA. Also found that the enzymatic product of PTGDS and prostaglandin D2 (PGD2) are raised in bald human scalp tissue. These results implicate that PGD2 might has a role in pathogenesis of AGA, thus suggest new receptor targets for its treatment.

Cetirizine, the active carboxylic acid metabolite of hydroxyzine, is a safe and selective second-generation histamine H1 receptor antagonist widely used in daily practice. It has anti-inflammatory properties and high specific affinity for histamine H1 receptors. Studies have shown cetirizine causes a significant reduction in both the inflammatory cell infiltrate and PGD2 production, and these effects are not related to its anti-H1 activity.

The oral administration of cetirizine is commonly leads to different systemic side effects as sedation, ocular dryness, tiredness and dry mouth. Thus, the topical formulation for cetirizine is expected to be a rational and effective tool for avoiding the oral side effects as well as better targeting, but unfortunately, no topical formulation of cetirizine is available in the market till date.

As the stratum corneum is the main barrier for the effective topical drug application, numerous attempts have been made to enhance topical drug delivery such as lipid nanocarriers (nano-transferosomes (NTF), follicular penetration, microbubbles and microneedles.

Rossi in 2018 evaluated for the first time in literature the tolerability and efficacy of topical cetirizine 1% lotion inpatients with AGA and claimed that topical cetirizine causes a significant improvement of the initial framework of AGA in both males and females and recommended further studies to allow better investigation for the role of cetirizine in AGA.

To the best of the investigators knowledge the use of topical cetirizine 1% gel has not yet been tried in the therapeutic management of Egyptian males with AGA.

ELIGIBILITY:
Inclusion Criteria:

1. Only males with Androgenetic Alopecia.
2. Age (18 - 50) years.
3. AGA grade II to VII according to Norwood-Hamilton classification

Exclusion Criteria:

1. Females with Androgentic Alopecia.
2. Previous history of sensitivity to Cetirizine.
3. Previous treatment for AGA in the last in the last 3 months
4. Chronic Systemic diseases as; hypotension, cardiac patients, renal failure or liver failure.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change of the hair density (follicles/cm²) | 6 months
  Improvement of the outcomes of treatment of androgenetic alopecia with Cetirizine 1% gel in comparison to Minoxidil 5% gel in terms of proportion of hair regrowth, the hair density (follicles/cm²) .

SECONDARY OUTCOMES:
Change of the hair diameter | 6 months
  Improvement of the vellus and terminal hair diameter <0.05 mm>

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Abd-ElMoez, Study Director — Professor of Dermatology, Venereology and Andrology, Faculty of Medicine, Assiut University
Locations (1):
- Assiut University, Asyut, Egypt